CLINICAL TRIAL: NCT06066385
Title: Suture Techniques to Reduce the Incidence of Incisional Hernia After Midline Laparotomy; Long-Term Follow-Up of the STITCH Trial
Brief Title: Suture Techniques to Reduce the Incidence of Incisional Hernia: LTFU STITCH Trial
Acronym: LTFU-STITCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Franciscus &Vlietland (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Rijnstate Hospital (Other); Spaarne Gasthuis (Other); Meander Medisch Centrum (Other); Red Cross Hospital Beverwijk (Other)
Responsible Party: Principal Investigator, Prof. dr. Pieter J Tanis, Prof.dr. P.J. Tanis, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9354; IIS WC-2022-06 (Other Grant/Funding Number: Ethicon Inc.); MEC 2022-0652 (Registry Identifier: METC)
Record Dates: First submitted 2023-09-01; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Surgery; Incisional Hernia; Wound Infection; Fascial Dehiscence; Pain; Quality of Life
Keywords: Surgery; Incisional Hernia; Wound Infection; Fascial Dehiscence; Pain; Quality of Life; Pathological Conditions, Anatomical; Infections; Postoperative Complications; Pathologic Processes
MeSH Terms: conditions — Incisional Hernia; Wound Infection; Pain; Pathological Conditions, Anatomical; Infections; Postoperative Complications; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: A Long-term follow-up with Outcome Assesor blinding of a parallel assigned double blinded (Participant, Investigator) Randomised Controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors of previous radiological imaging and imaging created during our Long-term follow up will be blinded to the assigned randomization arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small bites suturing technique of the abdominal wall during midline laparotomy (Experimental): In the experimental group of 288 patients the small bites technique was applied with bite widths of 0,5 cm and inter suture spacing of 0,5 cm with the use of PDS plus ll 2-0 single suture material with a 31 mm needle placed in the linea alba. In the small bites technique, twice as many stitches will be placed per sutured cm, with a smaller needle and thinner suture material.
  Interventions: Procedure: Small bites technique
- Large bites suturing technique of the abdominal wall during midline laparotomy (Active Comparator): As control the conventional large bites technique (mass closure) was applied with bites widths of 1 cm and inter-suture spacing of 1 cm with the use of PDS plus ll 1-0 double loop suture material with a 48 mm needle.
  Interventions: Procedure: Conventional large bites closure

INTERVENTIONS:
Procedure: Small bites technique — Closure of the fascia after midline laparotomy using a slowly resorbalbe 2.0 suture, with 0.5 cm bites, and 0.5 cm between the stitches, at least resulting in a 1:4 wound length:suture length ratio.
  Arms: Small bites suturing technique of the abdominal wall during midline laparotomy
Procedure: Conventional large bites closure — Closure of a midline laparotomy using a slowy resorbable thick suture (e.g. PDS loop) with large bites and large steps (>= 1 cm).
  Arms: Large bites suturing technique of the abdominal wall during midline laparotomy

SUMMARY:
Rationale: Incisional hernias (IH) are a frequent complication after abdominal surgery. Prevalence of an IH varies depending on the previous abdominal procedure but could be as high as 70% in high-risk patients after open surgery. To investigate different fascia closure techniques in the prevention of IHs, the STITCH trial (NCT01132209) was designed. The study compared two different closure techniques for closure of a midline incision in adult patients undergoing an elective abdominal laparotomy. Patients were randomly assigned to the intervention group (small bites 5 mm x 5 mm) or the control group (large bites 1 cm x 1 cm). The study showed that small bites are much more effective than large bites in the prevention of an incisional hernia when closing a midline incision.

So far, it has not been studied whether there is still a long-term difference in incidence of incisional hernia between the small bites and the large bites group.

Objective: The primary objective of this study is to determine the difference in incidence of IH between the small bites and the large bites group after 10 years of follow-up from time of randomization in the STITCH trial. The secondary objectives are to measure quality of life (QoL), body image and cosmetic results, and abdominal wall function through questionnaires and physical examination in those patients who are still alive.

DETAILED DESCRIPTION:
Rationale: Incisional hernias (IH) are a frequent complication after abdominal surgery. Prevalence of an IH varies depending on the previous abdominal procedure but could be as high as 70% in high-risk patients after open surgery. To investigate different fascia closure techniques in the prevention of IHs, the STITCH trial (NCT01132209) was designed, a randomized controlled trial in which 560 patients were included between October 2009 and March 2012. The study compared two different closure techniques for closure of a midline incision in adult patients undergoing an elective abdominal laparotomy. Patients were randomly assigned to the intervention group (small bites 5 mm x 5 mm) or the control group (large bites 1 cm x 1 cm). It showed that small bites are much more effective than large bites in the prevention of an incisional hernia when closing a midline incision.

So far, it has not been studied whether there is still a long-term difference in incidence of incisional hernia between the small bites and the large bites group.

Objective: The primary objective of this study study is to determine the difference in incidence of IH between the small bites and the large bites group after 10 years of follow-up from time of randomization in the STITCH trial. The secondary objectives are to measure quality of life (QoL), body image and cosmetic results, and abdominal wall function through questionnaires and physical examination in those patients who are still alive.

Study design: Assessment of long-term follow-up (10-13 years) of a randomized controlled multicenter study based on retrospective review of patient files and relevant imaging of the entire trial population, as well as questionnaires and physical and radiological examination of patient who are still alive.

Study population: Of the 560 included patients in the original STITCH trial, 545 completed the 1-year follow-up.

Intervention (if applicable): Not applicable. Main study parameters/endpoints: The primary outcome measure is the 10-year midline incisional hernia rate. The primary endpoint will be determined for the 545 patients of the original intention-to-treat population using Kaplan Meier analysis. In patients who died during follow-up, this will be evaluated by reviewing the available medical charts and radiological studies. CT-scans of the abdomen will be evaluated by the study-team. If CT imaging is not available, documented findings during physical examination by the relevant medical specialist will be considered. Patients being still alive with written informed consent to be contacted will be approached for their willingness to participate in this follow-up study, and after consent, we will reassess CT scans for an incisional hernia. All patients who are still alive and want to participate in this study will be asked to visit the hospital once for physical examination and an ultrasound of the abdominal wall.

Secondary outcome parameters include QoL and cosmetic outcome, Patients still alive with consent for participation will be sent the following questionnaires: MOS SF-36 and EQ-5D (QoL), Dresden Body Image Questionnaire (body image), Body Image Questionnaire (cosmesis), Hernia-Related Quality of Life Survey (abdominal wall function). Furthermore, readmission and surgical intervention rates related to midline IH will be determined for the entire study population.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Undergoing an ultrasound, physical examination and completing several questionnaires may be considered burdensome for the patient.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet the following criteria:

* Available signed informed consent form for the original STITCH trial of the patients who are still alive.
* Or if the patients has died, the medical records are reviewed.

A potential subject who meets the following criteria will be excluded from participation in this study:

- Patients that on the original informed consent form of the STITCH trial, checked the box that they did not want to be approached for future follow-up studies.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia occurrence (and timeto incisional hernia outcome). | Patients will have a follow-up of up to 12 years, with most patients having a follow-up between 10 and 12 years.
  Incisional hernia occurrence after operation clinical and/or radiological diagnosis.

SECONDARY OUTCOMES:
Quality of life of the patient. | Patients will have a follow-up of more than 10 years.
  Quality of life measured by MOS SF-36, ranging from 0 (worst) to 100 (best).
Quality of life of the patient. | Patients will have a follow-up of up to 12 years.
  Quality of life measured by and EQ-5D, ranging from 0 (worst) to 100 (best).
Body image. | Patients will have a follow-up of up to 12 years.
  Body image measured by Dresden Body Image Questionnaire (DBIQ), consisting of 35 questions that can be answered with a yes or no. This results in a range of 0 (worst) to 35 (best) points.
Cosmetic results, cosmesis. | Patients will have a follow-up of up to 12 years.
  Cosmetic results measured by Body Image Questionnaire (BIQ), consisting of 10 questions with a score ranging from 10 (worst) to 64 (best) points.
AWF. | Patients will have a follow-up of up to 12 years.
  Hernia-Related Quality of Life Survey (HerQLes), with 12 questions ranging from 12 (worst) to 72 (best) points.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter J Tanis, Principal Investigator — Erasmus Medical Center
Locations (9):
- Netherlands (9):
  - Erasmus MC, Rotterdam, South Holland
  - Meander Medical Center, Amersfoort
  - Rijnstate ziekenhuis, Arnhem
  - Red Cross Hospital, Beverwijk
  - Groene Hart Ziekenhuis, Gouda
  - Spaarne Gasthuis, Haarlem
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Prior Havenziekenhuis patients currently in the Erasmus MC, Rotterdam
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Original STITCH trial — https://pubmed.ncbi.nlm.nih.gov/26188742/

DOCUMENTS (1):
  • Study Protocol (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT06066385/Prot_000.pdf